CLINICAL TRIAL: NCT03093935
Title: StimRouter™ Neuromodulation System: Implanted Peripheral Nerve Stimulation for Pain Management When Treating Patients With Chronic Post-stroke Shoulder-pain
Brief Title: StimRouter™ for Pain Management in Post-stroke Shoulder Pain
Acronym: PSSP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of subject participation
Sponsor: Bioness Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STMR Pain 002 PSSP
Record Dates: First submitted 2017-03-18; First posted 2017-03-28 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Chronic Pain; Hemiplegic Shoulder Pain
Keywords: Post-Stroke; Neuromodulation; Axillary nerve; Peripheral Nerve Stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Cohort- Prospective, multi-center to collect population specific outcome measures in post-stroke patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- StimRouter Neuromodulation System (Experimental): All eligible patients who are enrolled in this study will be treated with StimRouter stimulation therapy as part of standard of care for the entire duration of the study (6 months) and observed for post-market population-specific data.
  Standard recommended stimulation parameters for post-stroke shoulder pain include settings to elicit sensory response (paresthesia) as well as motor response (muscle contraction).
  Interventions: Device: StimRouter Neuromodulation System

INTERVENTIONS:
Device: StimRouter Neuromodulation System — The StimRouter Neuromodulation System is indicated for pain management in adults who have severe intractable chronic pain of peripheral nerve origin, as an adjunct to other modes of therapy (e.g., medications). The StimRouter is not intended to treat pain in the craniofacial region.
  Other Names: StimRouter

SUMMARY:
StimRouter Neuromodulation System includes an implanted lead which provides peripheral nerve stimulation for chronic pain. Post-stroke shoulder pain patients will be the focus of this study. After meeting inclusion/exclusion criteria, approximately 50 enrolled patients will participate in the study through 6 months of follow-up. Various measures will be used to assess patient response to use of the device.

DETAILED DESCRIPTION:
Adults age 18 or over with severe intractable chronic shoulder pain subsequent to stroke will be included. Pain relief will be measured after using StimRouter stimulation therapy targeting the axillary nerve. Existing/pre-study pain medications must be either maintained, reduced throughout the trial.

Study Design is prospective, multi-center and will include 50 subjects The primary endpoint will be a clinically relevant pain reduction (30%) in pain score at 3 months after initiating stimulation in at least 50% of patients with no increase in pain medication.

Primary Outcomes: Reduction of average pain at rest measured by numeric scale (BPI-SF5)

Secondary Outcomes

1. Change in Worst Pain (BPI-SF3)
2. Least Pain & Pain Right Now (BPI - SF 4,6)
3. Patient Global Impression of Change (PGIC)
4. Patient Satisfaction questionnaire
5. Shoulder Q Data Collection Points

1) Baseline 2) Month 1 post-programming 3) Month 2 post-programming 4) Month 3 post-programming 5) Month 6 post-programming Data Analysis Analyses will be made to evaluate differences in outcomes compared to baseline measures, with primary endpoint at Month 3

* Standard statistical estimation and inference will be undertaken for the observed treatment effect.
* All adverse events will be tabulated by their frequencies and proportions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥18 years and confirmed diagnosis of stroke
* Competent to provide consent and comply with study requirements
* Minimum 3 months of severe chronic focal post-stroke shoulder pain
* Stable regimen of pain medications for >4 weeks prior to implant and willing to maintain equivalent dosage throughout the study
* A mean score of > 4 on the Brief Pain Inventory short form, question 3 (BPI-SF3)
* Capable and willing to follow all study-related procedures
* Able to tolerate surface stimulation as demonstrated by motor level response at shoulder

Exclusion Criteria:

* Patients who decline to provide written consent or to attend follow-up visits
* Shoulder pathology (e.g. rotator cuff tear, frozen shoulder etc) at target limb
* Evidence of a primary central or regional pain pattern inclusive of shoulder
* Diagnosed/confirmed shoulder dysfunction
* Botox or other neurolytic agent injections in last 3 months
* Any confounding neurologic conditions affecting the upper limb
* Evidence or history of skin infections
* History of adverse reactions to local anesthetics (e.g. lidocaine) or adhesives
* Patients who have an active systemic infection or are immunocompromised
* Patients who are pregnant, intend to become pregnant, are breastfeeding or of child-bearing potential and not practicing a medically-approved method of birth control
* Currently requiring or likely to require Magnetic Resonance Imaging (MRI) within the MRI exclusion zone defined as within 50cm of the iso-center or 16 cm of the MR coil as measured from the edge of the MRI coil.
* Any metallic implant in the immediate area intended for implant (e.g. TSR)
* Has demand-type cardiac pacemaker, defibrillator, or electrical nerve implant
* Potential need for diathermy at the implant site
* Potential need for therapeutic ultrasound at the implant site
* Patients who have already been implanted with StimRouter TM prior to study enrollment
* Presence of a documented condition or abnormality that could compromise the safety of the patient
* Life expectancy of less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) Change | Change from Baseline at Month 3
  The Brief Pain Inventory (BPI) form is a standard pain assessment tool based on a 0 to 10 scale. The Average Pain at Rest (BPI question number 5) score will be assessed at Baseline and approximately 3 months after programming (therapy start) to determine if there is a significant reduction in average pain with the addition of StimRouter TM treatment to standard of care.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) Change | Change from Baseline at Month 3
  Patient Global Impression of Change (PGIC) survey assesses perceived overall change in a combination of pain and life quality
Patient Satisfaction | Month 3
  Patient Satisfaction will be measured by a numeric (i.e., 1-5) rating scale (NRS)
Standardized Shoulder Questionnaire (Shoulder Q) Change | Change from Baseline at Month 3
  Change in difficulty level (on a scale from 0 to 3) or ability (yes/no) for completing normal day-to-day activities such as combing hair or lifting an 8 pound container to the shoulder level without bending the elbow, as measured by the Shoulder Q standardized questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Keith McBride, Study Chair — Bioness Inc
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No